CLINICAL TRIAL: NCT01044043
Title: Prevalence and Subjective Impairment of Quality of Life (QoL) Due to Dermatologic Diseases in Internal Medicine Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: University Hospital Zurich, Edouard Battegay, Switzerland: University of Zurich
Other Study IDs: PREV_DERM_INTMED
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Dermatologic Disease of Inpatients in Internal Medicine
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: clinical examination and quality of life questionnaire — clinical examination and quality of life questionnaire

SUMMARY:
This is a 3 months single centre clinical patient-oriented study to evaluate the prevalence and impairment in QOL of dermatologic diseases in patients hospitalised in internal medicine.

Up to 200 patients hospitalised at the division of internal medicine for any reason are going to be offered participation by a patient information form given to patients at the time of admission, as well as oral information about the study. Written informed consent will be obtained by the investigators after patients have had adequate time to consider their participation in the study.

Participating patients will be examined clinically for dermatologic pathologies at a single visit. In the case of signs of dermatologic disease, investigators are going to recommend further diagnostic procedures to the physician in charge and/or the referring physician, depending on the urgency of the suspected diagnosis. This procedure is meant to avoid giving referring physicians the impression that active patient acquisition for the department of Dermatology is an aim of this study. Diagnostic procedures that are performed upon suspicion of a specific dermatologic disease at the Division of Internal Medicine are going to be performed during the hospitalisation period. All other diagnostic or operative procedures are going to be advised to the referring physician.

Study participants are going to be interviewed by the investigators about impairment in QOL of their illnesses. Two separate questionnaires are going to be filled in by each participant. For measurement of general QOL, the widely used SF-12 questionnaire (8 questions) is going to be used. To measure specific impairment in QOL by dermatologic disease, participants are going to be asked to fill in the DLQI (Dermatology life quality index, 10 questions). Photographic documentation of specific identified lesions will be made and pictures stored exclusively in the secured electronic patient file (KISIM). Medication and all identified diseases will be noted. All diagnostically useful information is going to be recorded in the patient file and transmitted to the referring physician in the discharge letter.

ELIGIBILITY:
Inclusion criteria: Patients will be eligible for enrolment if they fulfil the following criteria:

1. Male or female patients, age ? 18 years of age and
2. Hospitalised at the Division of Internal Medicine, University Hospital Zurich
3. Patients must be able to give written informed consent before any trial-specific procedures are performed (see Section 12.2).

Exclusion criteria: Patients will be excluded from the study if they fulfill any of the following criteria:

1. Ability to communicate orally severely impaired due to any reason, namely illness or inability to speak German.
2. Terminal patients or other patients where participation in a visit with oral and physical examination would represent an unreasonable exertion.
3. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalance and subjective inpairment of quality of life due to dermatologic deseases in internal medicine patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland